CLINICAL TRIAL: NCT00713817
Title: A Multicentre, Open Label, Follow on Study to Assess the Maintenance of Effect, Tolerance and Safety of Sativex® in the Treatment of Subjects With Neuropathic Pain. This Will be Followed by a Randomised-withdrawal Phase (Part B) for a Subset of Patients
Brief Title: A Study to Determine the Maintenance of Effect After Long-term Treatment of Sativex® in Subjects With Neuropathic Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: GWCL0404 Part B
Record Dates: First submitted 2008-07-10; First posted 2008-07-11 (Estimated); Results first posted 2012-08-16 (Estimated); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Pain; Peripheral Neuropathy
Keywords: Pain; Peripheral Neuropathy
MeSH Terms: conditions — Pain; Peripheral Nervous System Diseases | interventions — nabiximols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sativex (Experimental)
  Interventions: Drug: Sativex®
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sativex® — Containing THC (27 mg/ml):CBD (25 mg/ml), in ethanol:propylene glycol (50:50) excipients, with peppermint oil (0.05%) flavoring. Maximum permitted dose was eight actuations in any three hour period and 24 actuations (THC 65 mg: CBD 60 mg) in 24 hours
  Other Names: GW-1000-02
  Arms: Sativex
Drug: Placebo — containing peppermint oil, 0.05% (v/v), quinoline yellow, 0.005% (w/v), sunset yellow, 0.0025% (w/v), in ethanol:propylene glycol (50:50) excipient
  Other Names: GW-4001-01
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the maintenance of effect after long-term treatment of Sativex® in subjects with neuropathic pain.

DETAILED DESCRIPTION:
A five week randomised-withdrawal phase (Part B) for a subset of subjects who took part in a 38 week, multicentre, open label (Part A) follow-on study to evaluate, the maintenance of effect of, the development of tolerance through exposure to, and safety of, Sativex® in the treatment of subjects with neuropathic pain. Subjects returned to the centre for an end of treatment visit at week 38 of Part A (Visit 5, Day 266), followed by Visits 5b (week 39), 5c (week 43) and an end of study visit took place 28 days after Visit 5c or withdrawal from the study.

ELIGIBILITY:
Inclusion Criteria:

* Had participated in GWCL0404, was currently ongoing in the study (i.e. still receiving GW-1000-02 treatment) and had completed the study up to Visit 5
* Had complied with all of the study requirements to-date, including the completion of the diary cards
* Had shown tolerability to the study medication in this study
* Ability (in the investigators opinion) and willingness to comply with all study requirements, including the completion of diary cards and study questionnaires

Exclusion Criteria:

* Had experienced or was currently experiencing any adverse events or untoward medical occurrences which, in the opinion of the investigator, would prevent them from safely participating in this phase of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2007-03; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Hoggart, MBBS, FRCA, Principal Investigator — Pain Management Research, Clinical Trials Unit, Netherwood House, Solihull Hospital
Locations (1):
- Pain Management Research, Clinical Trials Unit, Netherwood House, Solihull Hospital, Solihull, West Midlands, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Sativex: Contains Δ9 tetrahydrocannabinol (THC), 27 mg/ml: cannabidiol (CBD), 25 mg/ml delivered in 100 microlitre actuations by a pump action oromucosal spray. Maximum permitted dose was 24 actuations (THC 64.8 mg:CBD 60 mg) in 24 hours.
- Placebo: Contains no active drug but colourants and excipients. The maximum permitted dose was 24 actuations in any 24 hour period.
Period: Overall Study
Arm/Group | Sativex | Placebo
Started | 10 | 9
Completed | 10 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sativex | Placebo | Total
Number analyzed (Participants) | 10 | 9 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 8 | 18
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.7 (4.69) | 56.1 (10.33) | 53.8 (7.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 4 | 5 | 9
Region of Enrollment [Number; unit: participants]
  United Kingdom | 2 | 2 | 4
  Czech Republic | 8 | 7 | 15

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Daily Pain Severity on a 0-10 Numerical Rating Scale Score at the End of Treatment (Average of Last 7 Days Treatment)
Description: The pain severity Numerical Rating Scale was complete at the same time each day, i.e. bedtime in the evening. The patient was asked "on a scale of '0 to 10', please indicate the number that best describes your pain severity in the last 24 hours" where 0 = no pain and 10 = pain as bad as you can imagine. No pain relates to the time prior to the onset of neuropathic pain. A negative value indicates an improvement in pain score from baseline.
Time Frame: Day 0-35
Population: The efficacy analyses were conducted on data from all subjects who were randomised, received at least one dose of study medication and yielded on-treatment efficacy data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 10 | 9
units on a scale | 0.57 (1.06) | -0.49 (2.32)
Statistical Analysis 1: Comparison: Sativex vs Placebo; The two groups were compared using Analysis of Covariance (ANCOVA) with baseline severity as a covariate and study centre group and treatment group as factors. Due to the low power of the test for interaction the test was performed at the 10% level of significance and a 95% confidence interval (CI) was presented for the difference between treatments; Test type: Superiority or Other; p = 0.273, ANCOVA; Estimated mean treatment difference = 0.89, 95% CI 2-sided [-0.78 to 2.56]

2. Secondary Outcome: Change From Baseline Neuropathic Pain Score at the End of Treatment
Description: The Neuropathic Pain Scale score is the 0-100 sum of 10 individual pain scores (0-10 Numerical Rating Scale, 0= no pain to 10 = most pain imaginable). A negative change from baseline indicates an improvement in pain.
Time Frame: Day 7 to 35
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 10 | 9
units on a scale | 2.56 (5.57) | -2.06 (9.87)
Statistical Analysis 1: Comparison: Sativex vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.296, ANCOVA; Estimated mean treatment difference = 4.62, 95% CI 2-sided [-4.51 to 13.75]

3. Secondary Outcome: Number of Subjects Who Failed Treatment at the End of the Treatment Period
Description: Treatment failure was defined as follows:
  A. Premature termination of Part B (Randomised-Withdrawal) study medication. All subjects who did not complete at least 28 days on Part B (Randomised-Withdrawal) study medicationOr:
  B. An increase in pain, i.e. the mean pain 0-10 Numerical Rating Scale over seven consecutive days after Part B (Randomised-Withdrawal) randomisation had increased by at least 20% from the Part B (Randomised-Withdrawal) randomised treatment baseline.
Time Frame: Day 7 to time of last dose
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 10 | 9
participants | 5 | 4
Statistical Analysis 1: Comparison: Sativex vs Placebo; Time to treatment failure was analysed using Kaplan-Meier Survival analysis methodology. The difference in loss of response cumulative distribution function between treatments was assessed using the Hodges-Lehmann estimate; Test type: Superiority or Other; p = 0.826, Log Rank; Chi-square = 0.048

4. Secondary Outcome: Number of Subjects With More Than a 20% Loss of Response at the End of Treatment
Description: The percentage change from baseline in mean 0-10 Numerical Rating Scale pain score was calculated. The percentage changes from baseline were classified and the number of subjects with 20% or greater loss of response to treatment (i.e. percent increase from baseline ≥ 20%) is presented.
Time Frame: Day 0-35
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 10 | 9
participants | 3 | 2
Statistical Analysis 1: Comparison: Sativex vs Placebo; The difference in loss of response cumulative distribution functions between treatments was assessed using the Wilcoxon test with an estimate of the median difference between groups in response level (percent change from baseline) provided by the Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.54, Hodges-Lehmann; Estimated mean treatment difference = -7.14, 95% CI 2-sided [-39.7 to 9.62]

5. Secondary Outcome: Change From Baseline in Sleep Disruption 0-10 Numerical Rating Scale Score at the End of Treatment (Average of Last 7 Days Treatment)
Description: The sleep disruption Numerical Rating Scale was completed at the same time each day, i.e. bedtime in the evening. The patient was asked "on a scale of '0 to 10', please indicate how your pain disrupted your sleep last night?" where 0 = did not disrupt sleep and 10 = completely disrupted (unable to sleep at all). A negative value indicates an improvement in sleep disruption score from baseline.
Time Frame: Day 0-35
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 10 | 9
units on a scale | 0.24 (1.58) | 0.12 (0.97)
Statistical Analysis 1: Comparison: Sativex vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.902, ANCOVA; Estimate mean treatment difference = -0.08, 95% CI 2-sided [-1.45 to 1.29]

6. Secondary Outcome: Subject Global Impression of Change at the End of Treatment
Description: A 7-point Likert-type scale was used, with the question: 'Please assess the status of your nerve pain since entry into the study using the scale below' with the markers "very much improved, much improved, slightly improved, no change, slightly worse, much worse or very much worse". The number of subjects wo reported an improvement is presented.
Time Frame: Day 7 to 35
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 10 | 9
participants | 5 | 4
Statistical Analysis 1: Comparison: Sativex vs Placebo; The two treatment groups were compared using ordinal logistic regression and the proportional odds model. The model incorporated the parent Randomised Controlled Trials (RCTs). The interaction between treatment group and parent RCTs was investigated, but was dropped from the model if found to have little influence. The test was performed at the 10% significance level. The final model was then treatment group and parent RCTs, i.e. the treatment effect was adjusted for parent RCTs baseline; Test type: Superiority or Other; p = 0.603, Regression, Logistic; Odds Ratio (OR) = 1.557, 95% CI 2-sided [0.293 to 8.261]

7. Secondary Outcome: Incidence of Adverse Events as a Measure of Subject Safety
Description: The number of subjects who experienced an adverse event during the course of the study is presented.
Time Frame: Day 0 -35
Population: The safety analysis set comprised all subjects who received at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 10 | 9
participants | 3 | 2

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) occurring from the time of consent to post study follow up (63 days) were collected. All deaths and serious adverse events (SAEs) occurring within 28 days of the final dose of study medication were also collected.
Description: All AEs occurring during the study were reported on the running logs at the back of the study case report form.
Arm/Group | Sativex | Placebo
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/9
Other Adverse Events (participants affected / at risk) | 3/10 | 2/9
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sativex (N=10) | Placebo (N=9)
Headache (Nervous system disorders) | 2 | 0
Tremor (Nervous system disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Onychomycosis (Infections and infestations) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Weight decreased (Investigations) | 1 | 0
Stomach discomfort (Gastrointestinal disorders) | 0 | 1
Cataract (Eye disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GW will coordinate the dissemination of data from this study and may solicit input and assistance from the principal investigator. All publications, for example manuscripts, abstracts, oral/slide presentations or book chapters based on this study, must be submitted to GW for corporate review before release.